CLINICAL TRIAL: NCT02290925
Title: The Effect of a Biscuit Containing the Extract of Salacia Reticulata on Glycaemia in Patients With Type 2 Diabetes Mellitus Randomized Triple Blind Placebo Controlled Two Period Two Sequence Crossover Clinical Trial
Brief Title: The Effect of Biscuit Containing Kothala Himbutu on Blood Glucose in Patients With Diabetes. A Randomized Control Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rajarata University, Sri Lanka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RAJ-001
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: biscuit containing Salacia reticulate; randomised controlled trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — BAG 0177

STUDY DESIGN:
Intervention Model Description: Patients with diabetes were screened and Type I Diabetes was excluded. The minimum run-in period was eight weeks and if the variability of HbA1c is more than 20%, excluded, to exclude patients with fluctuating glycaemia. As this is a crossover trial some degree of stability of the glycemic control is necessary to prevent excessive variation of HbA1c interfering with the study outcome. Participants were randomized to receive the KH or placebo biscuit. Oral hypoglycemic was continued and adjusted. Participants consumed KH or placebo biscuit for a period of 3 months as mid-morning and afternoon snack. Subsequently in the washout period of 1 month the participants did not consumed any biscuits. After, crossing over they continued biscuits for another 3 months. HbA1c was done at recruitment, after run-in period, at 3 months and on completion of the study. When there was deterioration of the glycaemic control patient was prescribed insulin, and withdrawn from the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization code (A or B) was made using a computer and inserted in a sealed, serially numbered, opaque envelopes. Participants were given a serial number after run-in period. Assistant opened the envelope and assigned the patient to either biscuit A or B. The manufacturers held randomization code. Investigators, patients and those assessing the analysis were masked to the group outcome. Both Kothala Himbutu (KH) and placebo biscuits are identical in size, wrapped in same cover, and packed in identical boxes. The investigators tasted both biscuits and KH biscuits were slightly darker with the same taste. The study product is available in the market. Patients participating in the trial were asked about prior consumption of KH biscuits bought from the market (to exclude contamination). At the end of each period patients were asked whether they could assume the type of biscuit (KH biscuit or placebo) given to them and their preference for the type.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kothala Himbutu biscuit (Experimental): A biscuit containing Kothala Himbutu (Salacia reticulata) extract. This biscuit is available in the supermarkets. Four biscuits twice a day for 3 months.
  Interventions: Drug: Kothala Himbutu Biscuit
- placebo biscuit (Placebo Comparator): An identical biscuit without the herbal extract from Kothala Himbutu (Salacia reticulate)
  Interventions: Dietary Supplement: Placebo Biscuit

INTERVENTIONS:
Drug: Kothala Himbutu Biscuit — Kothala Himbutu biscuit (containing Salacia reticulata extract) as a snack. This herb has been used by traditional physicians to control blood sugar.
  Other Names: Biscuit contining Salacia reticulata extract; Kothala Himbutu Biscuit manufactured by Ceylon Biscuits Ltd; Munchee Kothala Himbutu biscuit
  Arms: Kothala Himbutu biscuit
Dietary Supplement: Placebo Biscuit — Placebo biscuit without the herbal extract of Kothala Himbutu (Salacia reticulate)
  Other Names: Biscuit; Munchee biscuit
  Arms: placebo biscuit

SUMMARY:
The investigators intend to conduct a triple blind randomized clinical trial to investigate the effect of a biscuit containing herbal extract, available in the market on the fasting blood sugar control in patients with diabetes mellitus and also to find out whether there are any side effects on other vital organs such as kidneys and liver.

DETAILED DESCRIPTION:
The effect of a biscuit containing the extract of Salacia reticulata (Kothala Himbutu) on the reduction of blood glucose levels in patients with Type 2 Diabetes Mellitus. A single center randomized triple blind placebo controlled two period two sequence crossover clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes for minimum period of 6 months
2. Aged between 30 and 65 years
3. Stable glycaemic control over the preceding 2-3 months. They will be initially selected from a range of HBA1C varying from 6.5 - 14 and the individual subject should not have a variation of >20% between the previous HBA1C and the HBA1C done at the commencement of the study

Exclusion Criteria:

1. Chronic kidney disease with estimated Glomerular filtration rate less than 30ml/hour
2. Severe valvular heart disease or heart failure.
3. Those on Insulin therapy
4. Severe liver disease (AST > 10 X times the upper limit)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeesha Wickramasinghe, BSc, Study Director — Faculty of Medicine & Allied Sciences, Rajarata University of Sri Lanka
Locations (1):
- Teaching Hospital Anuradhapura, Anuradhapura, North Central Province, Sri Lanka

IPD SHARING:
Plan to Share IPD: Yes
Individual Patient Data (IPD) will be available for researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 10 years after end of the study (March 2019)
Access Criteria: Any qualified researcher should submit the protocol and get the ERC clearence from institutional IRB (Ethics Review Committee, Faculty of Medicine & Allied Science, Rajarata University of Sri Lanka). After that they need to come to an written agreement with the researchers to analyze the data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment carried out in medical clinic, Teaching Hospital anuradhapura
Pre-assignment Details: Run-in period was 8 weeks and if the variability of the HbA1c is more than 20%, participants were excluded. This was done to exclude patients with fluctuating glycaemia.
  Wash out for 1 month after 1st period of giving treatment for 3 months. After the wash out patients are crossed over for the other biscuit given for another three months
Groups:
- Placebo Biscuit First and Then Kothala Himbutu Biscuit: (Description of the placebo biscuit, and the Kothala Himbutu biscuit is described in the other arm)) An identical placebo biscuit without the herbal extract from Kothala Himbutu (Salacia reticulate). Given as same as the Kothala Himbutu biscuit and manufactured by the same manufacturer.
- Kothala Himbutu Biscuit First and Then Placebo Biscuit: A biscuit containing Kothala Himbutu (Salacia reticulata) extract. This biscuit is available in the supermarkets. Four biscuits twice a day as a mid morning and a mid afternoon snack for 3 months. Dry bark of the Salacia reticulate plant (210kg) is boiled repeatedly with water and evaporated to 210 liters of extract containing 10.5kg of dried extract (Herbal drug to extract ratio 1:1). The 100g of biscuit mixture are blended with 1.042ml of the aqueous extract. The raw material was authenticated by thin layer chromatography finger print analysis by the Industrial Technology Institute, Colombo. The energy, carbohydrate and fiber content of the study and the placebo biscuits are identical. The KH biscuit contained 447.21kcal of energy, 10.42g of protein, 13.97g of fat (6.29g saturated), 69.95g of carbohydrates (less than 0.10g of sugar), 7.53g of dietary fiber and 979mg of sodium per 100g. Glycaemic index of the KH biscuit was 30 and the placebo biscuit was 56.
Period: First Period of Three Months
Arm/Group | Placebo Biscuit First and Then Kothala Himbutu Biscuit | Kothala Himbutu Biscuit First and Then Placebo Biscuit
Started | 62 | 71
Completed | 58 | 69
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 1 | 0
Not completed — Insulin Started | 1 | 1
Period: Second Period of 3 Months
Arm/Group | Placebo Biscuit First and Then Kothala Himbutu Biscuit | Kothala Himbutu Biscuit First and Then Placebo Biscuit
Started | 58 | 69
Completed | 57 | 65
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 3
Not completed — insulin started | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Biscuit First Then Kothala Himbutu Biscuit Group: first given placebo biscuit for three months and after wash out period of one month given Kothala Himbutu biscuit (extract of Salacia reticulata) for three moths
- Kothala Himbutu First Then Placebo Biscuit Group: first given Kothala Himbutu biscuit (extract of Salacia reticulata) for three months and after wash out period of one month given placebo biscuit for three moths
- Total: Total of all reporting groups
Arm/Group | Placebo Biscuit First Then Kothala Himbutu Biscuit Group | Kothala Himbutu First Then Placebo Biscuit Group | Total
Number analyzed (Participants) | 62 | 71 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 62 | 71 | 133
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (8.4) | 50.7 (7.1) | 50.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 51 | 93
  Male | 20 | 20 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 62 | 71 | 133
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sri Lanka | 62 | 71 | 133
Glycosylated Haemoglobin [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] — Blood samples were analyzed at a centrally accredited lab and HBA1c was measured using ion exchange high performance liquid chromatography standardized to NGSP
  percentage of glycosylated haemoglobin | 8.45 (1.40) | 8.65 (1.44) | 8.56 (1.42)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin
Description: HBA1c were analyzed at a centrally accredited lab using ion exchange high performance liquid chromatography standardized to NGSP
Time Frame: After 3 months and after 7 months (there is one month wash over period as this is a cross over trial)
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- Kothala Himbutu Biscuit First Then Placebo Biscuit Group: first given Kothala Himbutu biscuit (extract of Salacia reticulata) for three months and after wash out period of one month given placebo biscuit for three moths
Arm/Group | Placebo Biscuit First Then Kothala Himbutu Biscuit Group | Kothala Himbutu Biscuit First Then Placebo Biscuit Group
Number analyzed (Participants) | 62 | 71
percentage of glycosylated hemoglobin
  After period 1(3 months) | 8.36 (0.19) | 8.16 (0.20)
  After period 2 (trial end-7 months) | 8.23 (0.21) | 8.53 (0.21)
Statistical Analysis 1: Comparison: Placebo Biscuit First Then Kothala Himbutu Biscuit Group vs Kothala Himbutu Biscuit First Then Placebo Biscuit Group; Test type: Other — general linear model (GLM) with repeated measures; Mean Difference (Net) = 0.25 — Box's M tests was used. Mauchly's test was used to verify that the error covariance matrix of the orthonormalized-transformed dependent variables is proportional to an identity matrix; We used intention to treat analysis. Since the missing data were more than 5%, we examined the dataset to determine whether it shows "missing completely at random" (MCAR) "not missing at random (NMAR)" or "data missing at random" (MAR). A sensitivity analysis was done to determine whether multiple imputations are required. It included complete case analysis, best-worst case and worst best case scenario with group mean±1SD

2. Secondary Outcome: Liver Adverse Effects
Description: liver functions are described in the table below with higher liver enzymes suggesting injury to the liver.
Time Frame: Baseline, after 3 months, and after 7 months
Population: adverse events analysis was only people who have completed or accessible for analysis. this was not a intention to treat analysis
Measure: Mean (Full Range); unit: International Units per Liter
Groups:
- Kothala Himbutu Biscuit First and the Placebo Biscuit Group: first given Kothala Himbutu biscuit (extract of Salacia reticulata) for three months and after wash out period of one month given placebo biscuit for three moths
Arm/Group | Placebo Biscuit First Then Kothala Himbutu Biscuit Group | Kothala Himbutu Biscuit First and the Placebo Biscuit Group
Number analyzed (Participants) | 62 | 71
International Units per Liter
  ALT (IU/L) at baseline | 38 [12 to 95] | 37 [9 to 129]
  ALT (IU/L) after 3 months: number analyzed (Participants) | 58 | 69
  ALT (IU/L) after 3 months | 39 [12 to 124] | 36 [11 to 111]
  ALT (IU/L) after 7 months: number analyzed (Participants) | 57 | 65
  ALT (IU/L) after 7 months | 37 [11 to 110] | 34 [12 to 90]
  AST (IU/L) at baseline | 28 [11 to 97] | 28 [11 to 111]
  AST (IU/L) after 3 months: number analyzed (Participants) | 58 | 69
  AST (IU/L) after 3 months | 28 [11 to 132] | 26 [10 to 73]
  AST (IU/L) after 7 months: number analyzed (Participants) | 57 | 65
  AST (IU/L) after 7 months | 27 [12 to 90] | 24 [10 to 55]

3. Secondary Outcome: Renal Adverse Effects -1
Description: Renal functions are described in the table below with Lower estimated Glomerular Filtration Rate (eGFR) suggesting injury to the kidney.
Time Frame: baseline, after 3 months and after 7 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: milliliters/minute/1.73m^2
Arm/Group | Placebo Biscuit First Then Kothala Himbutu Biscuit Group | Kothala Himbutu Biscuit First Then Placebo Biscuit Group
Number analyzed (Participants) | 62 | 71
milliliters/minute/1.73m^2
  eGFR (ml/min/1.73m^2) at baseline | 77.1 [41 to 90] | 76.0 [41 to 90]
  eGFR (ml/min/1.73m^2) after 3 months: number analyzed (Participants) | 58 | 69
  eGFR (ml/min/1.73m^2) after 3 months | 75.0 [39 to 90] | 75.0 [41 to 90]
  eGFR (ml/min/1.73m^2) after 7 months: number analyzed (Participants) | 57 | 65
  eGFR (ml/min/1.73m^2) after 7 months | 75.0 [41 to 90] | 76 [41 to 90]

4. Secondary Outcome: Renal Adverse Effects - 2
Description: Renal functions are described in the table below with higher serum creatinine suggesting injury to the kidney.
Time Frame: Baseline, after 3 months, and after 7 months
Population: as for outcome 2
Measure: Mean (Full Range); unit: milligrams per deciliter
Arm/Group | Placebo Biscuit First Then Kothala Himbutu Biscuit Group | Kothala Himbutu Biscuit First Then Placebo Biscuit Group
Number analyzed (Participants) | 62 | 71
milligrams per deciliter
  Serum creatinine (mg/dL) at baseline | 0.94 [0.04 to 1.84] | 0.94 [0.10 to 1.47]
  Serum creatinine (mg/dL) after 3 months: number analyzed (Participants) | 58 | 69
  Serum creatinine (mg/dL) after 3 months | 0.98 [0.70 to 1.97] | 0.96 [0.62 to 1.70]
  Serum creatinine (mg/dL) after 7 months: number analyzed (Participants) | 57 | 65
  Serum creatinine (mg/dL) after 7 months | 0.97 [0.60 to 1.80] | 0.93 [0.61 to 1.39]

ADVERSE EVENTS:
Time Frame: seven months
Description: Renal or urinary disorder and Hepato-biliary disorder were systematically collected. All other adverse events were monitored.
Groups:
- Placebo Biscuit Group: Adverse events are reported "per intervention" (participants consuming placebo biscuits are presented here). Separate Arms/Groups reflect all participants who received each intervention during the study.
- Kothala Himbutu Biscuit Group: Adverse events are reported "per intervention" (participants consuming Kothala Himbutu biscuits are presented here). Separate Arms/Groups reflect all participants who received each intervention during the study.
Arm/Group | Placebo Biscuit Group | Kothala Himbutu Biscuit Group
All-Cause Mortality (participants affected / at risk) | 1/131 | 0/129
Serious Adverse Events (participants affected / at risk) | 1/131 | 0/129
Other Adverse Events (participants affected / at risk) | 0/131 | 0/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Biscuit Group (N=131) | Kothala Himbutu Biscuit Group (N=129)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — death due to pneumonia

LIMITATIONS AND CAVEATS:
Withdrawing patients needing insulin from the trial compromised the pragmatic nature of the RCT. Blinding of the patients may have been affected because of the slightly different taste and darker nature of the KH biscuit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT02290925/Prot_SAP_000.pdf